CLINICAL TRIAL: NCT00292175
Title: Randomised,Controlled Trial of Narrow Band Imaging With Magnification (NBI) Versus White Light Endoscopy for Dysplasia Detection in Ulcerative Colitis Surveillance
Brief Title: NBI With Magnification for Dysplasia Detection in Ulcerative Colitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London North West Healthcare NHS Trust (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 06/NBI2/10
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-09

CONDITIONS: Ulcerative Colitis
Keywords: colonoscopy, narrow band imaging (NBI), ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Narrow Band Imaging; Colonoscopy

INTERVENTIONS:
Procedure: Narrow Band Imaging
Procedure: colonoscopy

SUMMARY:
The purpose of the study is to determine whether a new colonoscopic viewing technique called narrow band imaging (NBI) helps doctors detect more patients with at leat one pre-cancerous area (dysplasia associated lession or mass, MALMs) than conventional colonoscopy using white light alone.

DETAILED DESCRIPTION:
Colorectal cancer is the second commonest cause of cancer death. Patients with colitis have a substantially increased risk of death from colorectal cancer which increases with lenght of time the patient has had colitis. This can be as high as a 30% chance of colorectal cancer after 30 years of colitis. Colonoscopic surveillance of colitis patients has been shown to reduce the risk of colorectal cancer and allow detection at an earlier stage, but even with meticulous examination, some precancerous lesions or cancers are missed.

Precancerous lesions in colitis are difficult to see and endoscopist have used spraying dye on the lining of the bowel (chromoendoscopy) successfully to improve detection of abnormal areas: however this is time consuming and requires extra time and equipment and despite the benefits seen in multiple studies is not widely used in routine clinical practice in the UK.

Narrow band imaging (NBI) is a technique that relies on light filters to improve contrast for the smallest blood vessels in the bowel lining which shows up precancerous areas as they have a richer vascular network. It is sometimes described as "digital chromoendoscopy" as the images produced are similar to chromoendoscopy, but it is much simpler and quicker to use. With magnification it allows assessment of the fine mucosal surface pattern (pit pattern) of lesion which allows and assessment of their likelihood of being precancerous. Autofluorescence endoscopy uses short wavelength light and light filters to produce a false colour image of the bowel lining where polyps stand out. These techniques have been used with some success in the oesophagus and stomach but little work is available for the colon.

We aim to see if NBI with magnification is better that standard colonoscopy for detecting precancerous areas. This is likely as it produces images similar to chromoendoscopy which is already shown to help. If a potentially precancerous area is found we will use other types of endoscopy, particularly NBI autofluorescence to see if these techniques are helpful for discriminating between pre-cancerous and non pre-cancerous areas

ELIGIBILITY:
Inclusion Criteria:

* petients with colitis who meet surveillance criteria
* patients over 18 years of age

Exclusion Criteria:

* pregnant patients
* unable or unwilling to give informed consent
* patients with severe active colitis who would be unsafe to endoscope

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2006-02

PRIMARY OUTCOMES:
Effectiveness of NBI versus Light endoscopy

SECONDARY OUTCOMES:
Are more precancerous lessions found in total with NBI?
Are more advanced precancerous lesions found with NBI?
Are more patients found with more that one precancerous lesion with NBI?
How Many lessions are successfully completely removed via the endoscope?

CONTACTS AND LOCATIONS:
Overall Officials: Brian Saunders, MD, FRCP, Principal Investigator — London North West Healthcare NHS Trust
Locations (2):
- United Kingdom (2):
  - North West London Hospitals NHS Trust - St Mark's, London, Middlesex
  - Nottingham Univesrity Hospitals NHS Trust, Queen's Medical Centre, Nottingham